CLINICAL TRIAL: NCT03669770
Title: Ultrasound Classification and Grading of Lipohypertrophy and Its Impact on Glucose Variability in Type 1 Diabetes: The TITANIC Studies.
Brief Title: Ultrasound Classification and Grading of Lipohypertrophy and Its Impact on Glucose Variability in Type 1 Diabetes
Acronym: TITANIC
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 217187
Record Dates: First submitted 2018-06-28; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2017-08

CONDITIONS: Lipohypertrophy; Type 1 Diabetes Mellitus
Keywords: Lipohypertrophy; Type 1 Diabetes Mellitus; Ultrasound; Glucose variability; Glycaemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will use ultrasound to characterise lipohypertrophy(LH) and assess the impact of LH on glucose variability in adults with type 1 diabetes. LH is a condition that occurs with repeated exposure to insulin at injection sites, resulting in the development of subcutaneous fatty lumps that impede the absorption of insulin. LH can lead to glucose variability, increased risk of severe hypoglycaemia and diabetes distress. In the long term it can therefore lead to increased risk of diabetes complications and increased insulin costs.

DETAILED DESCRIPTION:
This is an observational study using ultrasound (US) to assess and characterise lipohypertrophy (LH) with a sub-study to assess the impact of LH on glucose variability in a case-crossover study.

The study aim is to assess LH using ultrasound and its impact on glucose variability.

The objectives of the study are:

1. To use ultrasound to characterise (appearance, location, mass, and distribution) LH tissue in participants with T1DM injecting insulin.
2. To develop a standard operating procedure for using US to assess LH.
3. To develop a grading system to evaluate LH using US.
4. To investigate the relationship between the observed LH and glucose variability, glycaemic control, and/or severe hypoglycaemia.
5. To assess quality of life, diabetes distress, and insulin treatment satisfaction after moving to a new injection site and being alerted to the existence of LH.
6. To learn more about how people living with type 1 manage their injection sites.

Study design:

All patients attending the diabetes clinics in Guys and St Thomas' Foundation Trust with type 1 diabetes for more than three years and thought to have LH will be offered the opportunity to participate in the study. Those testing their glucose four or more times a day and with a standard deviation of their mean glucose greater than 4mmols, will be offered to participate in the case-crossover arm of the study; a sub-study, which forms a students doctoral studies.

All participants will be asked to give demographic details and medical history. They will be asked to complete a series of questionnaires about their injection technique, diabetes distress, insulin treatment satisfaction and quality of life. All participants will have a baseline glycated haemoglobin taken, and for those in the case-crossover study an additional 1,5-anhydroglucitol and insulin antibody tests done. The case-crossover study with then be fitted with a continuous glucose monitoring (CGM) device to record their glucose variability for the following six days. They will then return for the US assessment of their injection sites and digital palpation; while all other participants in the characterisation study only, will have had this done at the first visit. All participants will be advised as to where they have LH and where they can inject to avoid LH and after five weeks in the case of the case-crossover study return for a second CGM of six days, and then all participant return after six weeks for the final visit.

At this visit they will complete the questionnaires for a second time and a short exit interview will be conduct to gather information on their experience of injecting into a LH free site and injecting insulin. The glycated haemoglobin will be repeated and for the case-crossover study another 1,5-anhydroglucitol will be taken. Finally, the participants will have a session with a diabetes specialist nurse, who will advise them on maintaining a stable glucose level and refer on as appropriate to their diabetes team.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Type 1 Diabetes Mellitus (T1DM)
* Age> 20 years
* Taking multiple daily injections ≥4 per/day
* Diagnosed T1DM and using insulin for >3 years
* Using the same insulin type and delivery method for past 6 months
* Ability to speak and read English

Case-crossover study:

* Glucose variability with a Standard deviation ≥4mmol/l of mean glucose in the previous four weeks
* ≥4 blood glucose tests per/day

Exclusion Criteria:

* Age <20 years
* Type 2 diabetes or Gestational diabetes mellitus (GDM)
* Have a condition or receiving therapies, other than insulin, associated with lipodystrophies
* Have another medical condition or take medicines that may influence blood glucose control (including: currently active cancer; uncontrolled endocrine disorder; eating disorders; celiac disease; and cystic fibrosis)
* Have a serious medical or mental health condition that impairs full engagement in the research
* Using other injectable treatments in diabetes such as growth hormone or glucagon like peptide-1.
* Using Continuous Subcutaneous Insulin Infusion (CSII)
* Not undertaking blood glucose tests ≥4 tests per day
* Unable to speak English or unable to give consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All T1DM patients attending the diabetes clinics in GSTFT thought to have have LH and fitting the above criteria.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Changes in Glucose variability between baseline and follow-up | 6 weeks
  Glucose variability will be measured using the standard deviation of the mean glucose measured at visit 1 and the last visit. For the case-crossover study the data will be taken from the CGM recording and the other participants with their own self-monitoring of glucose measurements.
Changes in Glycaemic control between baseline and follow-up | 6 Weeks
  Glycaemic control will be assessed in all participants using glycated haemoglobin at first clinical outpatient appointment and at six weeks. In addition, participants at the case-crossover study will have a 1, 5 anhydroglucitol taken at study visit 1 and at six weeks.

OTHER OUTCOMES:
Time patient spends in the hypoglycaemic/ hyperglycaemic state | 6 weeks
  Time spend in the hypoglycaemic (Low blood glucose) and hyperglycaemic (High blood glucose) range as indicated by Continuous Glucose Monitoring data.
Various glucose variability measures | 6 Weeks
  standard deviation(SD) of mean glucose; coefficient of variation (CV); mean amplitude of glycaemic excursion(MAGE); continuous overall net glycaemic action(CONGA-n); and mean of daily differences(MODD). These will be identified from the Continuous Glucose Monitoring data.
Changes of the Insulin dosage requirements | 6 Weeks
  Total daily dose (proportion of basal and bolus insulin) at baseline and follow-up
Diabetes Distress | 6 Weeks
  Diabetes distress will be measured using the 17-item diabetes distress scale at baseline and follow-up (Polonsky et al. 2005, Fisher et al. 2008).
Insulin Treatment Satisfaction | 6 Weeks
  Insulin Treatment Satisfaction Questionnaire (ITSQ) at baseline and follow-up (Anderson et al. 2004)
Health-related quality of life | 6 Weeks
  Health related quality of life be assessed with the EuroQol EQ-5D-5L questionnaire at baseline and follow-up (Herdman et al. 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Angus Forbes, Professor, Study Director — King's College London
Locations (1):
- Florence Nightingale Faculty of Nursing, Midwifery & Palliative Care, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No